CLINICAL TRIAL: NCT05570799
Title: Effect of Using Gamification and Augmented Reality in Mechanical Ventilation Teaching on Nursing Students' Knowledge, Motivation, and Self-Efficacy: A Randomized Controlled Trial
Brief Title: Gamification and Augmented Reality in Mechanical Ventilation Teaching for Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Sahar Younes, Assistant professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AR and Game based learning
Record Dates: First submitted 2022-10-01; First posted 2022-10-07 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Gamification; Augmented Reality
Keywords: Gamification; Augmented reality; knowledge; self-Efficacy; motivation; Mechanical Ventilation Teaching; Critical Care Nursing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No augmented reality or Kahoot game-based learning group (traditional lectures group)
- Experimental group (Experimental): Augmented reality learning and Kahoot game group
  Interventions: Other: Augmented Reality and Kahoot game learning

INTERVENTIONS:
Other: Augmented Reality and Kahoot game learning — * An augmented reality (AR) mobile application with image based will be used by the participants in the experimental group.
  * Also, students will participate in Kahoot game. Students will participate in the game using their own devices by going to https://kahoot on their phones and entering their password and password.
  Arms: Experimental group

SUMMARY:
This study is designed to examine the effect of using gamification and augmented reality in mechanical ventilation teaching on Critical Care Nursing students' knowledge, self-efficacy, and motivation.

DETAILED DESCRIPTION:
A pretest-posttest, prospective, randomized controlled trial will be conducted. Random assignment will place participants in either the experimental group using augmented reality games or the control group using traditional lectures (control group).

1. Preparation of Augmented Reality Models

   * Mechanical ventilator handout will be developed by the authors. This handout will be including images of physiology of respiration, mechanical ventilator machines, ventilator graphs, and ventilator settings.
   * An augmented reality (AR) mobile application with image based AR will be used by the participants in the experimental group. The three-dimensional (3D) virtual models and images will be shown in the AR handout, and the participants could display the objects on the mobile screen with the use of a marker on the page of the AR handout using the camera in the mobile app.
2. Preparation of Kahoot Game

   * A teacher account was constructed on Kahoot after signing up at "https://kahoot.com".
   * A Kahoot quiz with 20 multiple-choice questions and pictures will be constructed at "https://create.kahoot". Only one correct option will be possible for each of the 20 questions.
   * When a quiz is created and opened in "Kahoot".
   * The students access to Kahoot within the classical game mode (Player vs Player "1:1 Devices").
   * A typical session of Kahoot involves 200 students playing the game.
   * Once each teaching unit is completed, students will be asked to actively participate in the classroom using Kahoot.
   * Once all of the players' names have appeared on the screen, the teacher presses "START" to begin the quiz.
   * Students' responses and the scores' calculation will be automatically stored in the database.
   * After the test is finished, a report of the results will be created and made available for download to the researcher.

Data Collection Procedure

The study will be conducted between October 20, 2022 and December 30, 2022.

* The students in experimental group received a 30 minutes augmented reality games training for mechanical ventilator using a 3D images and videos.
* The control group will be learned with the traditional materials in which the teacher will give online lectures regarding the mechanical ventilation utilizing PowerPoint presentation through Microsoft Teams platform.
* The self-administered questionnaires of knowledge, self-efficacy and motivation survey will take 15 minutes to complete for each participant via an online form. The pretest for both groups will be administered on the first day of the study, and the post-test will be administered immediately after and after three weeks of the intervention.
* Three weeks after the baseline measurements, knowledge, self-efficacy and Motivation Survey will be assessed again.

ELIGIBILITY:
Inclusion Criteria:

* Third-year nursing students enrolled in the course of Critical Care Nursing (I) for the first time;
* Smartphone owners and users; those who have internet access;
* Those who understood the goal and nature of the study and voluntarily agreed to participate

Exclusion Criteria:

* Prior experience in mechanical ventilation
* Refusal to participation

Ages: 19 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 410 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation knowledge test | through study completion, an average of 4 weeks
  It is a self-administered questionnaire that will be developed and used to assess students. The knowledge questionnaire contained 20 multiple choice questions
Self-efficacy | through study completion, an average of 4 weeks
  It was created using a five-step nursing process: clinical nursing skill assessment, problem diagnosis, clinical nursing skill preparation, skills performance, and evaluation.
Motivation Survey | through study completion, an average of 4 weeks
  Learning motivation was evaluated using a tool based on the Instructional Materials Motivation Scale (IMMS). The IMMS will be utilized to measure motivation-related problems in the self-directed learning of students.

SECONDARY OUTCOMES:
Students' opinions | through study completion, an average of 4 weeks
  To investigate students' opinions on game based learning strategy, a survey consisting of 4 items was conducted at the end of the retention test: ''To what extent were you motivated to learn? To what extent did you gain knowledge on mechanical ventilation? Did you find the mechanical ventilation game or lecture interesting? Did you enjoy the mechanical ventilation game or lecture?'' The first 2 items are rated on a 5-point Likert-scale from 1 (strongly disagree) to 5 (strongly agree), the last 2 items are answered with yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Y Othman, Ass. Prof., Principal Investigator — Faculty of Nursing, Damanhour University
Locations (1):
- Faculty of nursing, Damanhūr, Behira, Egypt

REFERENCES:
- [Background] Barsom EZ, Graafland M, Schijven MP. Systematic review on the effectiveness of augmented reality applications in medical training. Surg Endosc. 2016 Oct;30(10):4174-83. doi: 10.1007/s00464-016-4800-6. Epub 2016 Feb 23. PMID 26905573
- [Background] Muangpoon T, Haghighi Osgouei R, Escobar-Castillejos D, Kontovounisios C, Bello F. Augmented Reality System for Digital Rectal Examination Training and Assessment: System Validation. J Med Internet Res. 2020 Aug 13;22(8):e18637. doi: 10.2196/18637. PMID 32788146
- [Background] Felszeghy S, Pasonen-Seppanen S, Koskela A, Nieminen P, Harkonen K, Paldanius KMA, Gabbouj S, Ketola K, Hiltunen M, Lundin M, Haapaniemi T, Sointu E, Bauman EB, Gilbert GE, Morton D, Mahonen A. Using online game-based platforms to improve student performance and engagement in histology teaching. BMC Med Educ. 2019 Jul 22;19(1):273. doi: 10.1186/s12909-019-1701-0. PMID 31331319
- [Derived] Othman SY, Ghallab E, Eltaybani S, Mohamed AM. Effect of using gamification and augmented reality in mechanical ventilation unit of critical care nursing on nurse students' knowledge, motivation, and self-efficacy: A randomized controlled trial. Nurse Educ Today. 2024 Nov;142:106329. doi: 10.1016/j.nedt.2024.106329. Epub 2024 Aug 5. PMID 39116661